CLINICAL TRIAL: NCT04861090
Title: Retrospective, Observational Chart Review Study Evaluating Clinical Effectiveness and Disease/Treatment Management Among Patients Who Initiated Long-term Prophylaxis With Takhzyro® in a Real-world Setting
Brief Title: A Study in Teenagers and Adults With Hereditary Angioedema (HAE) Type I or Type II Who Use Lanadelumab as Long-Term Prophylaxis
Acronym: INTEGRATED
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4006; MACS-2020-081002 (Other: Takeda)
Record Dates: First submitted 2021-04-19; First posted 2021-04-27 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Hereditary Angioedema: Participants with HAE type I or type II who had initiated long-term prophylaxis (LTP) treatment with lanadelumab which was administered every two weeks (Q2W) or every four weeks (Q4W) or every six weeks (Q6W) or every eight weeks (Q8W) in accordance to Summary of Product Characteristics (SmPC), during a routine clinical setting will be followed up to 38 months.

SUMMARY:
The main aims of this study are to learn how many people with HAE Type I or Type II are attack-free when treated with lanadelumab in real life. This includes the number of people that are attack-free when lanadelumab is given every 2 and every 4 weeks.

This study is about collecting existing data only; participants will not receive lanadelumab as part of this study. No new information will be collected during this study. Only data already available at the participant's doctor's office will be reviewed and collected for this study.

Participants do not need to visit their doctor in addition to their normal visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged >= 12 years at the time of the last documented HAE attack in the eligibility period.
* Participant has a physician-confirmed diagnosis (or confirmation in medical records) of HAE type I or type II.
* Participant had initiated LTP with lanadelumab during the eligibility period.
* Participant provides informed consent or assent prior to the initiation of any study procedures (where required by local regulations).

Exclusion Criteria:

* Participant was enrolled in a therapeutic investigational drug or device trial during the observation period.
* Participant without documented HAE attacks in the pre-index period and/or without available participant diary or systematic documentation of HAE attacks in the medical records during the post index period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult or adolescent participants (aged greater than or equal to [>=] 12 years) with HAE type I or type II who initiated LTP treatment with lanadelumab within a routine clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Are Free of Hereditary Angioedema (HAE) Attacks Treated With Lanadelumab | Up to Month 12
  Percentage of participants who are free of HAE attacks will be reported. A HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Percentage of Participants Who Are Free of HAE Attacks Treated With Lanadelumab Administered Every Two Weeks | Up to Month 12
  Percentage of participants who are free of HAE attacks treated with lanadelumab which was administered every two weeks will be reported.
Percentage of Participants Who Are Free of HAE Attacks Treated With Lanadelumab Administered Every Four Weeks | Up to Month 12
  Percentage of participants who are free of HAE attacks treated with lanadelumab which was administered every four weeks will be reported.

SECONDARY OUTCOMES:
Percentage of Participants With Specific HAE Attack Occurrence | Up to Month 12
  Percentage of participants with specific HAE attack occurrence (e.g. attacks of specific localization, attacks requiring on-demand medication, life-threatening attacks) will be reported.
Percentage of Participants Who are Free of HAE Attacks Relative to Prior Treatment | Up to Month 12
  Percentage of participants who are free of HAE attacks relative to prior treatment (e.g. prior prophylaxis treatment or on-demand medications) among participants treated with lanadelumab will be reported.
Number of Participants Characterized With Every Four Weeks Adjustment | Every 4 weeks from start of treatment (Up to Month 12)
  Number of participants will be characterized with every four weeks adjustment (e.g. weight, age, duration of disease, history of life-threating attacks, length of attack-free interval during lanadelumab treatment) will be reported.
Number of Participants Characterized Based on Primary Reasons for Down Titration | Up to Month 12
  Number of participants will be characterized based on primary reasons for down titration will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- Austria (3):
  - LKH-Universitätsklinikum Klinikum Graz, Graz
  - Kepler Universitätsklinikum Linz, Linz
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
- France (7):
  - CHU de Grenoble, Grenoble
  - CHRU Lille, Lille
  - Groupement Hospitalier Edouard Herriot, Lyon
  - CHU Montpellier - Hôpital St Eloi, Montpellier
  - Hôtel Dieu de Paris Hospital, Paris
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Universitaire Hopitaux de Rouen, Rouen
- Germany (7):
  - Charitè Campus Mitte, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hanover
  - Hämophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
  - Klinikum rechts der Isa der Technischen Universitaet Muenchen, Munich
  - Universitatsklinikum Munster, Münster
  - Universitätsklinikum Ulm, Ulm
- Greece (3):
  - Navy Hospital of Athens, Athens
  - Laiko General Hospital of Athens, Athens
  - University General Hospital of Larissa, Larissa

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Magerl M, Bouillet L, Martinez-Saguer I, Gavini F, Bent-Ennakhil N, Sayegh L, Andresen I. Real-World Effectiveness of Lanadelumab in Hereditary Angioedema: Multicountry INTEGRATED Observational Study. J Allergy Clin Immunol Pract. 2025 Feb;13(2):378-387.e2. doi: 10.1016/j.jaip.2024.12.008. Epub 2024 Dec 17. PMID 39701274
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/608ac7aef89629001e47b4e8